CLINICAL TRIAL: NCT03087331
Title: An Evaluation of the Effect of Community-based Pharmacist Intervention on Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21092
Record Dates: First submitted 2016-05-10; First posted 2017-03-22 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Medication Review; Restraint, Physical; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacist intervention (Experimental): Within the pharmacist intervention arm, pharmacists will do medication reviews, assessment, recommendations, education.
  Interventions: Other: medication reviews, assessment, recommendations, education.

INTERVENTIONS:
Other: medication reviews, assessment, recommendations, education.

SUMMARY:
This is a prospective, pre post, pilot cohort study to be conducted in patients with chronic pain, which is defined as pain that lasts beyond 3 months. To accomplish the primary and secondary objectives of the study, three phrases will be designed and completed during three months

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of community-based pharmacist interventions on the quality of life of patients with chronic pain as determined by self-reported pain levels using an established scoring system. Participating pharmacists will enroll chronic pain patients from their normal practice to receive a consultation, which consists of an assessment of their current pain, a medication review, and education about their condition. Based on the information provided by the patient, the pharmacist will prepare a care plan, contact the patient's prescriber, and, in conjunction with the prescriber, implement the plan to help relieve their pain. Follow-up assessments will be done after 2 weeks, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or older
2. Baseline average pain intensity using Brief Pain Inventory is 6 or higher
3. Ambulatory and able to attend the intervention
4. Complaining of pain for 3 months or longer

Exclusion Criteria:

1. Patients with malignant or cancer pain
2. Patients who are unable to communicate in English
3. Non-ambulatory and unable to attend the intervention at the participating site
4. Unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity change | baseline, 2 weeks follow-up, 3 months follow-up
  Pain intensity will be measured with Brief Pain Inventory pain intensity subscale, and will be measured 3 times in total

SECONDARY OUTCOMES:
Pain interference | baseline, 2 weeks follow-up, 3 months follow-up
  Pain interference will be measured with Brief Pain Inventory pain interference subscale, and will be measured 3 times in total
Quality of life change | baseline, 3 months follow-up
  quality of life will be measured using Short Form-36, and will be measured twice in total.

OTHER OUTCOMES:
patient adherence | 2 weeks follow-up and 3 months follow-up
  Patient adherence will be measured using Morisky medication adherence scale-8, and will be measured at 2 weeks and 3 months follow-up.The Morisky medication adherence scale-8 will be used as supplementary data to further elucidate potential factors behind the observed outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Chang, Study Director — University of Waterloo
Locations (1):
- The PharmaShoppe, Kitchener, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No